CLINICAL TRIAL: NCT00966771
Title: Preventing Future Pregnancy After Choosing the Copper IUD vs. Oral Levonorgestrel for Emergency Contraception
Brief Title: The Copper T380A IUD vs. Oral Levonorgestrel for Emergency Contraception
Acronym: IUD EC
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Society of Family Planning (Other)
Responsible Party: Principal Investigator, David Turok, Clinical Assistant Professor, University of Utah
Other Study IDs: 30937; 1R21HD063028-01A1 (NIH)
Record Dates: First submitted 2009-08-25; First posted 2009-08-27 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2016-10

CONDITIONS: Pregnancy
Keywords: contraception; emergency contraception; pregnancy prevention after unprotected intercourse
MeSH Terms: interventions — Levonorgestrel

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- IUD: Women presenting for emergency contraception who select the copper IUD
  Interventions: Drug: Copper T380 IUD
- Oral levonorgestrel: Women presenting for emergency contraception who select oral levonorgestrel
  Interventions: Drug: Oral levonorgestrel

INTERVENTIONS:
Drug: Copper T380 IUD — copper T 380 IUD
  Other Names: Paragard IUD
  Groups: IUD
Drug: Oral levonorgestrel — 1.5 mg
  Other Names: Plan B
  Groups: Oral levonorgestrel

SUMMARY:
The purpose of this study is to see if women presenting for emergency contraception (EC) and choose the copper intrauterine device (IUD) will have fewer unplanned pregnancies in the next year compared to women who choose oral levonorgestrel for EC. The study will also compare use of an effective method of contraception in the year after they received EC.

DETAILED DESCRIPTION:
All women presenting to 2 Planned Parenthood Association of Utah clinics in Salt Lake City will be offered participation in this study. Women will select either the copper IUD or oral levonorgestrel for EC. The primary outcome is unplanned pregnancy in the year following presentation for EC.

Secondary outcomes include use of an effective method of contraception over the next year, abortions, repeat use of EC, number of days to first bleeding episode and duration of that bleeding episode, use of a barrier method to prevent sexually transmitted infections, patient satisfaction with the chosen method of EC and contraception. Participants selecting the IUD will be assessed for IUD expulsion, perforation, and removal.

ELIGIBILITY:
Inclusion Criteria:

* Women 18-30 years old,
* in need of emergency contraception (had unprotected intercourse within 120 hours),
* willing to give consent for participation in research,
* willing to comply with study requirements, and
* accessible by telephone.

Participants selecting the IUD need to identify themselves as desiring long-term contraception.

Exclusion Criteria:

* Current pregnancy
* Had pelvic inflammatory disease or septic abortion within the past 3 months or had gonorrhea or chlamydia infection in the last 60 days
* Current behavior suggesting a high risk for pelvic inflammatory disease
* Allergy to copper or Wilson's disease (for participants selecting the copper IUD) or allergy to levonorgestrel (for participants selecting oral levonorgestrel)
* Abnormalities of the uterus that distort the uterine cavity
* Mucopurulent cervicitis
* A previously placed IUD that has not been removed
* Genital bleeding of an unknown etiology
* Ovarian, cervical, or endometrial cancer
* Small uterine cavity (< 6cm)

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women presenting to family planning clinics for emergency contraception
Sampling Method: Non-Probability Sample
Enrollment: 548 (Actual)
Dates: Start 2009-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Unplanned pregnancy | within 12 months of presenting for EC

SECONDARY OUTCOMES:
Use of an effective method of contraception in the year following use of emergency contraception. | 12 months
IUD expulsion, removal or perforation | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: David Turok, MD, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - Planned Parenthood Association of Utah Salt Lake City Clinic, Salt Lake City, Utah
  - Planned Parenthood Association of Utah, West Valley City Clinic, West Valley City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Royer PA, Turok DK, Sanders JN, Saltzman HM. Choice of Emergency Contraceptive and Decision Making Regarding Subsequent Unintended Pregnancy. J Womens Health (Larchmt). 2016 Oct;25(10):1038-1043. doi: 10.1089/jwh.2015.5625. Epub 2016 Mar 31. PMID 27032057
- [Derived] Torres LN, Turok DK, Sanders JN, Jacobson JC, Dermish AI, Ward K. We should really keep in touch: predictors of the ability to maintain contact with contraception clinical trial participants over 12 months. Contraception. 2014 Dec;90(6):575-80. doi: 10.1016/j.contraception.2014.07.013. Epub 2014 Aug 1. PMID 25242443